CLINICAL TRIAL: NCT07123532
Title: PREVALENCE OF SCAPULAR DYSKINESIS AMONG PHYSICAL THERAPY PRACTITIONERS AN EPIDEMIOLOGICAL STUDY
Brief Title: PREVALENCE OF SCAPULAR DYSKINESIS
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reda Abd Elaziz Ibrahim Abdo, general preactitioner, Cairo University
Other Study IDs: P.T.REC/012/005755
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Shoulder Pain
Keywords: Muscle Weakness; Scapular Dyskinesis
MeSH Terms: conditions — Shoulder Pain; Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- o Group A:: 27-31 years
- o Group B:: Above 31-36 years
- o Group C:: Above 36-40 years

SUMMARY:
Objective:

This study will aim to determine the prevalence of scapular dyskinesis (SD) among Egyptian physical therapy practitioners and will explore associated epidemiological factors, including age, sex, BMI, shoulder and neck symptoms, and scapular stabilizer muscle strength.

Design:

A cross-sectional observational study will be conducted, including 121 licensed Egyptian physical therapists aged 27 to 40 years. Participants will be divided into three age-based groups.

Methods:

Each participant will undergo a clinical examination for SD using the Scapular Dyskinesis Test (SDT) and the Lateral Scapular Slide Test (LSST). Pain intensity will be assessed using the Visual Analog Scale (VAS), and musculoskeletal symptoms will be recorded using the Nordic Musculoskeletal Questionnaire (NMQ). Shoulder range of motion and the strength of scapular stabilizer muscles (serratus anterior, middle, and lower trapezius) will also be evaluated. Statistical analysis will include Chi-square tests and one-way ANOVA at a significance level of p < 0.05.

DETAILED DESCRIPTION:
This study will be a cross-sectional observational study designed to investigate the prevalence of scapular dyskinesis (SD) among physical therapy practitioners and to explore associated epidemiological factors. The study will be conducted between October 2024 and January 2025. Ethical approval will be obtained from the Research Ethics Committee of the Faculty of Physical Therapy, Cairo University (P.T.REC/012/005755).

Participants

Sample Size: The sample size will be calculated using SPSS for Windows, version 25, with 80% power at α = 0.05 level using a one-sample t-test. The generated sample size will be 121 physical therapy practitioners.

Selection Criteria:

Inclusion Criteria:

Licensed physical therapy practitioners actively working in clinical settings (Soliño et al., 2024).

Age between 27 and 40 years (Jeong & Kim, 2023).

Minimum of one year of clinical experience or exposure to physical activity (Jeong & Kim, 2023).

No current shoulder pain or symptoms at the time of assessment (Soliño et al., 2024).

Willingness to participate and provide informed consent.

Exclusion Criteria:

Acute shoulder or neck injury within the last month (Jeong & Kim, 2023).

History of upper body orthopedic surgery (Jeong & Kim, 2023).

Known neurological or musculoskeletal disorders affecting shoulder mechanics (Burn et al., 2016).

Participation in overhead or collision sports with high scapular loading (Burn et al., 2016).

Inability to complete assessment procedures due to physical limitations (Soliño et al., 2024).

Subgroups: Participants will be divided into three age-based groups:

Group A: 27-31 years

Group B: Above 31-36 years

Group C: Above 36-40 years

Instrumentation

Body Mass Index (BMI): Weight and height will be measured using calibrated scales, and BMI will be calculated as body mass (kg) / height² (m²). A cutoff of ≥30 kg/m² will be considered obese (Romero et al., 2008).

Scapular Dyskinesis Test (SDT): Will be used to visually assess scapular movement patterns during repeated shoulder flexion and abduction with light weights (Plummer et al., 2017).

Lateral Scapular Slide Test (LSST): Will assess scapular position by measuring the distance from the scapula's inferior angle to the nearest spinous process in different arm positions. A side-to-side difference >1.5 cm will indicate asymmetry (Curtis et al., 2006).

Digital Goniometer: Will be used to assess shoulder range of motion (ROM) with alignment to anatomical landmarks (Correll et al., 2018; Norkin & White, 2016).

Visual Analog Scale (VAS): Will be used to measure pain intensity on a 10 cm line from 0 (no pain) to 10 (worst pain) (Begum et al., 2019).

Nordic Musculoskeletal Questionnaire (NMQ): An Arabic-adapted version will be used to assess musculoskeletal symptoms in specific body regions (Aldhabi et al., 2024).

Manual Muscle Testing (MMT): Strength testing of middle trapezius, lower trapezius, and serratus anterior will be conducted using the Oxford scale (Vijian et al., 2023).

Assessment Procedures

Personal Data: Name, age, sex, weight, and height will be recorded. Informed consent will be obtained from all participants.

BMI Calculation: Weight and height will be measured, and BMI will be computed using the standard formula (Abrantes et al., 2002).

Pain Assessment (VAS): Participants will mark their pain level on a 10 cm visual analog scale.

SDT: Participants will perform repeated shoulder flexion and abduction; abnormal scapular motion will be recorded as "yes" and normal as "no" (Jayasinghe, 2018).

LSST: Bilateral measurements will be taken in different arm positions; >1.5 cm difference will be considered abnormal (Jayasinghe, 2018).

Shoulder ROM Measurement: A digital goniometer will be used; the joint will be positioned and stabilized before measurement (Norkin & White, 2016).

NMQ Administration: A self-administered questionnaire will address demographic, biomechanical, psychological, and environmental factors (Smith et al., 2006).

MMT: Strength of scapular stabilizers will be graded on the Oxford scale; only grade 5 will be included in analysis to avoid confounding.

Glenohumeral Joint Assessment: Passive ROM will be evaluated for pain response and end-feel categorization (Norkin & White, 2016).

Statistical Analysis Data will be expressed as mean ± SD. The Shapiro-Wilk test will be used for normality testing. ANOVA will be applied to compare characteristics among the three subgroups, and the Chi-square test will be used to compare categorical variables. Statistical analysis will be performed using SPSS version 20 (SPSS Inc., Chicago, IL, USA), with significance set at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

Licensed physical therapy practitioners actively working in clinical settings (Soliño et al., 2024).

Age between 27 and 40 years (Jeong & Kim, 2023).

Minimum of one year of clinical experience or exposure to physical activity (Jeong & Kim, 2023).

No current shoulder pain or symptoms at the time of assessment (Soliño et al., 2024).

Willingness to participate and provide informed consent.

Exclusion Criteria:

Acute shoulder or neck injury within the last month (Jeong & Kim, 2023).

History of upper body orthopedic surgery (Jeong & Kim, 2023).

Known neurological or musculoskeletal disorders affecting shoulder mechanics (Burn et al., 2016).

Participation in overhead or collision sports with high scapular loading (Burn et al., 2016).

Inability to complete assessment procedures due to physical limitations (Soliño et al., 2024).

Ages: 27 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This cross-sectional observational study will investigate the prevalence of scapular dyskinesis (SD) among licensed physical therapy practitioners in Egypt and will explore associated epidemiological factors. The study will be conducted between October 2024 and January 2025 after obtaining ethical approval from the Research Ethics Committee, Faculty of Physical Therapy, Cairo University (P.T.REC/012/005755).
  A total of 121 participants will be recruited based on a sample size calculation with 80% power at α = 0.05 (one-sample t-test). Eligible participants will be aged 27-40 years, actively working in clinical settings, with at least one year of clinical experience or exposure to physical activity, and free from current shoulder symptoms. Exclusion criteria will include recent acute shoulder/neck injury, history of upper body orthopedic surgery, neurological or musculoskeletal disorders affecting shoulder mechanics, high scapular-loading sports participation, and inability to complete
Sampling Method: Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11-28 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Scapular Dyskinesis | At baseline (single assessment session).
  Determined by the proportion of participants diagnosed with abnormal scapular movement patterns using the Scapular Dyskinesis Test (SDT) and Lateral Scapular Slide Test (LSST).
  Measurement Method:
  SDT: Observation of scapular motion during repeated shoulder flexion and abduction with light weights. Abnormal motion recorded as "Yes," normal as "No."
  LSST: Measurement of distance from scapular inferior angle to the nearest spinous process in different arm positions; >1.5 cm side-to-side difference indicates dyskinesis.

SECONDARY OUTCOMES:
Shoulder Range of Motion (ROM) | At baseline.
  Measurement of active and passive ROM of the shoulder joint in degrees.
  Measurement Method: Digital goniometer aligned with anatomical landmarks (Norkin & White, 2016).
Scapular Stabilizer Muscle Strength | At baseline.
  Strength of the serratus anterior, middle trapezius, and lower trapezius.
  Measurement Method: Manual Muscle Testing (MMT) using Oxford scale; grade 5 only included in statistical analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt